CLINICAL TRIAL: NCT06346977
Title: A Prospective Study on the Diagnosis of Leptomeningeal Metastasis and the Monitoring of Intrathecal Chemotherapy Efficacy in NSCLC Based on Proteomics
Brief Title: Diagnosis of Leptomeningeal Metastasis and the Monitoring of Intrathecal Chemotherapy Efficacy in NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaorong Dong, Professor/Chief Physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: DTO-20231214
Record Dates: First submitted 2024-03-27; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Diagnosis
MeSH Terms: conditions — Disease | interventions — Pemetrexed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In Part One of the study, plasma samples (1 mL) were collected from NLM group participants at the time of initial diagnosis, when they presented with no clinical symptoms or radiological evidence of meningeal metastasis. For LM group subjects, both plasma (1 mL) and cerebrospinal fluid (2 mL) were obtained within two weeks prior to receiving intrathecal chemotherapy.
  In Part Two, plasma and CSF were gathered from cohort subjects at three time points: within two weeks before intrathecal chemotherapy (baseline), at T0 (24 hours post-injection), and at T28 (28 days post-injection), with 1 mL of plasma and 2 mL of CSF collected at each instance. Plasma was acquired through venipuncture, while CSF was extracted via lumbar puncture. All collected samples were earmarked for proteomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LM group;: Leptomeningeal Metastasis Group
  Interventions: Drug: Pemetrexed
- NLM group: Non-Leptomeningeal Metastasis Group

INTERVENTIONS:
Drug: Pemetrexed — Intrathecal injection of pemetrexed
  Groups: LM group;

SUMMARY:
Non-small cell lung cancer (NSCLC), occupying a disquieting position as the second most prevalent and deadliest neoplasm worldwide, afflicts an estimated 30% of its patients with intracranial metastatic spread. Among these, leptomeningeal metastasis (LM) is an exceptionally surreptitious and perilous manifestation, often evading timely and accurate diagnosis. The clinical landscape is further complicated by the presence of patients who, due to various reasons, are unable to undergo lumbar puncture, a procedure crucial for the investigation of LM. Moreover, even when cerebrospinal fluid (CSF) analysis via conventional cytological and immunohistochemical methods is attempted, a definitive diagnosis of LM may remain elusive in a subset of cases.

Intrathecal chemotherapy, particularly via the administration of pemetrexed, which has demonstrated both notable efficacy and an acceptable safety profile when delivered directly into the cerebrospinal space, constitutes a cornerstone of treatment for NSCLC-LM. Despite its importance, the lack of robust, validated biomarkers to gauge the therapeutic response to such interventions represents a significant knowledge gap. This deficit is compounded by the inherent challenges associated with CSF samples, including their limited availability and the suboptimal sensitivity and high resource demands of current ctDNA assessment techniques.

To address these pressing diagnostic and monitoring needs in NSCLC-LM management, the investigator proposes a forward-looking, non-interventional clinical study harnessing the power of cutting-edge proteomic technologies. These platforms, characterized by their high throughput, exquisite sensitivity, and minimal sample volume requirements, offer a promising avenue for elucidating the intricacies of chemotherapy response in intrathecal therapy. The study aims to provide valuable insights into improving diagnostic accuracy for LM in NSCLC patients and to establish a more rigorous framework for assessing treatment efficacy in individuals undergoing intrathecal chemotherapy, ultimately contributing to enhanced patient care and personalized therapeutic strategies.

DETAILED DESCRIPTION:
The research is structured into two distinct phases. In the inaugural segment, the investigator plans to assemble a comprehensive dataset by procuring plasma or cerebrospinal fluid (CSF) samples from 30 individuals presenting with confirmed CSF positivity for LM, juxtaposed against an equal number of advanced NSCLC cases manifesting neither clinical signs nor radiographic indicators of meningeal involvement. These biological materials will be subjected to rigorous proteomic interrogation, with the overarching goal of discerning distinctive proteomic signatures that can accurately discriminate between NSCLC patients with and without LM.

In the subsequent phase, the study's focus shifts to therapeutic response monitoring. Maintaining the same cohort of CSF-positive NSCLC-LM patients initially recruited in Phase One, the researcher will systematically collect plasma and CSF samples at critical junctures during their treatment trajectory: specifically, within the two-week period preceding intrathecal chemotherapy initiation (establishing a baseline), immediately following the intervention at T0 (24 hours post-administration), and at the T28 milestone (28 days post-injection). Simultaneously, meticulous documentation of each patient's treatment response, disease progression dynamics, and overall survival metrics will be meticulously compiled. This concerted effort is designed to harness the power of proteomics in providing a real-time, molecular snapshot of chemotherapy effectiveness, thereby offering invaluable insights into the therapeutic efficacy of intrathecal chemotherapy in the context of NSCLC-LM management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Histologically or cytologically confirmed diagnosis of NSCLC, stage IV according to the 8th edition of the International Association for the Study of Lung Cancer (IASLC) TNM Staging Manual
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2
* At least one lesion meeting the target lesion (TL) criteria of RECIST 1.1 at baseline. Must have imaging documentation of pretreatment tumor assessment by CT or MRI scan performed within 28 days before treatment initiation
* No prior intrathecal chemotherapy

Exclusion Criteria:

* History of allogeneic organ transplantation
* Active or documented history of autoimmune or inflammatory disorders (including inflammatory bowel disease [such as colitis or Crohn's disease], diverticulitis [except diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener's syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, pituitary itis, uveitis, etc.])
* Active history of primary immunodeficiency
* History of another malignancy within the past 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed primary non-small cell lung cancer (NSCLC), are staged as IV according to the 8th edition of the American Joint Committee on Cancer (AJCC) staging system.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to a maximum of 36 months.
  From the date of intrathecal drug administration until the date of first documented disease progression or death due to any cause, whichever occurs first, with an assessment period up to a maximum of 36 months.

SECONDARY OUTCOMES:
Overall survival (OS) | up to a maximum of 36 months.
  From the date of intrathecal drug administration until the date of death due to any cause, whichever occurs first, with an assessment period up to a maximum of 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Ping, Dr., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No